CLINICAL TRIAL: NCT04624802
Title: The Effect of Maternal Exercise on Anxiety During Normal Pregnancy：a Randomized Controlled Trial
Brief Title: Maternal Exercise and Antenatal Anxiety
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shenzhen Second People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20200601031-FS01
Record Dates: First submitted 2020-10-11; First posted 2020-11-12 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Anxiety
Keywords: anxiety; pregnancy; exercise
MeSH Terms: conditions — Anxiety Disorders; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- maternal exercise training group (Experimental): Pregnant women in experimental group are invited to participate in 16 exercise weekly classes for 40 min including 15 min aerobic exercise，10 min relaxation exercise, and 15 min aerobic exercise, from week 16 to week 32 of gestation, and receive antenatal care and examination regularly.
  Interventions: Behavioral: maternal exercise
- antenatal care group (No Intervention): Pregnant women in antenatal care group receive antenatal care and examination regularly.

INTERVENTIONS:
Behavioral: maternal exercise — The maternal exercise is broadly practiced by pregnant women in China. It is designed by a team led by Shen Shanmei, a professor of Maternity Exercises at Department of Obstetrics and Gynecology of First Hospital in Korea.
  Arms: maternal exercise training group

SUMMARY:
This is a randomized controlled trial study. We evaluate effectiveness of maternal exercise on anxiety during normal pregnancy compared to those who receive antenatal care regularly. We plan to recruit 220 healthy pregnant women over the age of 18 in Shenzhen and to use a standard maternal exercise from Korea as intervention.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who are over 18 years old and confirmed to be pregnant in Shenzhen Dapeng New District.

Exclusion Criteria:

* 1.pregnant women who have accepted maternal exercise training (at least twice a week in last month);2.pregnant women who have orthopedics, cardiovascular or mental diseases; 3.pregnant women who have or had any condition as follows:miscarriage more than two times,premature delivery,placenta previa,fetal dysplasia, low weight before pregnancy (BMI <17.5),polycyesis,preeclampsia,premature rupture of membranes,Uterine growth retardation,cervical/ligation,repeated vaginal bleeding,anemia or diabetes; 4.the gestational age is less than 12 weeks or more than 16 weeks;5.received psychotherapy or psychotropic medication within 6 months before the study;6.can not participate in regular inspections.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2020-11-10 (Estimated); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline of State Anxiety at 32 Weeks of Gestation | The participants are examined between 12 and 16 weeks of gestation (baseline visit) and at gestation week 32 (after the intervention).
  We use state anxiety subscale of State-Trait Anxiety Inventory (STAI) as the measure of anxiety severity. The STAI comprises two-self report scales for measuring two distinct anxiety concepts, the State anxiety and Trait anxiety. Both scales contain 20 statements that ask the respondent to describe how she feels at a particular moment (state anxiety) or how she generally feels (trait anxiety). State anxiety is conceptualized as a transitory emotional state, where as trait anxiety refers to relatively stable individual differences in proneness to anxiety. The respondents are required to rate themselves on a four point likert scale 'not at all' to 'very much so on' various anxiety related symptoms which they experience in the past weeks for the state scale or how they generally feel for the trait scale. STAI is widely used and has been shown to have high reliability and validity with a Cronbach's alpha of 0.88 and 0.83 for state (STAI-I) and trait anxiety (STAI-II) respectively.

SECONDARY OUTCOMES:
Change from Baseline of Depressive Symptom at 32 Weeks of Gestation | The participants are examined between 12 and 16 weeks of gestation (baseline visit) and at gestation week 32 (after the intervention).
  We use Beck Depression Inventory second edition (BDI-Ⅱ) as the measure of depressive symptom severity. The BDI-II is a 21-item self-report measure of common depressive symptoms. Each item has four possible responses, and higher total scores are indicative of a greater number and severity of depressive symptoms. Scores ranging from 0 to 13 indicate minimal/no symptoms, 14-19 indicate mild depression, 20-28 indicate moderate depression, and 29-63 indicate severe depression.
Change from Baseline of Pain at 32 Weeks of Gestation | The participants are examined between 12 and 16 weeks of gestation (baseline visit) and at gestation week 32 (after the intervention).
  We use Brief Pain Inventory (BPI) as the measure of the severity of pain. The pain intensity section of the BPI is composed by four items that are scored from 0 (no pain) to 10 (worst pain), while the functional interference section is composed by seven items that are scored from 1 (no interference with activities of daily living) to 10 (total interference). The severity index is calculated on the basis of the mean of the four pain intensity items, and interference index is calculated from the mean of the seven pain interference items.